CLINICAL TRIAL: NCT05364125
Title: Effect of Olfactory Training on Olfactory Dysfunction Patients in Hong Kong Population
Brief Title: Olfactory Training on Smell Dysfunction Patients in HK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Fergus Wong Kai Chuen, Associate Consultant, Pamela Youde Nethersole Eastern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OlfactoryTrainingHKRCT
Record Dates: First submitted 2022-04-14; First posted 2022-05-06 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Olfaction Disorders; Smell Disorders; Anosmia; Hyposmia; Olfactory Impairment; Smell Loss; Smell Dysfunction
MeSH Terms: conditions — Olfaction Disorders; Anosmia | interventions — Olfactory Training

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Randomly assigned by computer into treatment group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): Olfactory training by neurological chemosensory stimulation using aromatic substances delivered via diffusers. Four aromatic substances will be used. Each substance will be given for 20 seconds sequentially, providing a total of 80 seconds of olfactory stimulation three times per day for 3 months.
  Interventions: Other: Olfactory Training
- Control arm (Placebo Comparator): Same diffuser will be given to control group. All of the four essential oils will be replaced by normal saline using the same packing. Same treatment regime of 20 seconds for each diffuser three times per day for 3 months will be instructed to control group patients.
  Interventions: Other: Control

INTERVENTIONS:
Other: Olfactory Training — Four aromatic substances will be used (Citrus limon, Eucalyptus radiata, Pelargonium graveolens, Juniperus virginiana)
  Arms: Treatment arm
Other: Control — Normal Saline will be used
  Arms: Control arm

SUMMARY:
* Causes of olfactory dysfunction can be classified into conductive and sensorineural causes.
* Conductive causes are mainly due to structural nasal problem, which can be treated by nasal surgery
* Sensorineural causes included post-infection, post-head injury, post Head and Neck irradiation and other central nervous system diseases.
* Olfactory Training is well established treatment for sensorineural olfactory dysfunction in foreign countries.
* Olfactory Training by neurological chemosensory stimulation using aromatic substances delivered via electronic portable aromatic rehabilitation (EPAR) diffuser was proved to be effective treatment in COVID-19 related olfactory dysfunction in recent Hong Kong study.
* However, there is a lack of local study on the effect of Olfactory Training in other non-COVID-19 sensorineural causes of olfactory dysfunction in Hong Kong population.

DETAILED DESCRIPTION:
Design Prospective double-blinded randomized control trial.

Study Period 1/7/2022 - 30/6/2024 for case recruitment.

Suitable patient will be recruited. Informed consent will be signed. Objective smell assessment will be done using the University of Pennsylvania Smell Identification Test (UPSIT) and Butanol Threshold Test (BTT). Subjective quality of life score will be obtained by Sino-Nasal Outcome Test (SNOT-22). Subjective smell and taste assessment will be assessed by Visual Analogue Scale (VAS). Patient will be randomized into treatment group and control group using computer generated list by an independent nursing staff. Doctors and the patients will be blinded during the study.

ELIGIBILITY:
Inclusion Criteria:

* Olfactory dysfunction > 6 months and < 5 years

Exclusion Criteria:

* History of significant head injury (fracture, ICH)
* History of brain surgery
* History of nasal surgery
* Active nasal disease
* Active neurological disease
* Poor premorbid status/ non-communicable patients
* Mentally incompetent patients
* <18 years' old
* Pregnancy
* Hypersensitivity to the aromatic substance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Olfactory threshold changes after olfactory training after 3 months | 3 months after starting smell training
  Parameter:
  Olfactory threshold using Butanol Threshold Test (BTT)
Olfactory identification score changes after olfactory training after 3 months | 3 months after starting smell training
  Parameter:
  Olfactory identification using Smell Identification Test (UPSIT)
Quality of life changes after olfactory training after 3 months | 3 months after starting smell training
  Parameter:
  Subjective quality of life score using Sino-Nasal Outcome Test (SNOT-22)
Taste and smell changes after olfactory training after 3 months | 3 months after starting smell training
  Parameter:
  Subjective smell and taste assessment using Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Chuen Fergus Wong, FRCSEd(ORL), Principal Investigator — Pamela Youde Nethersole Eastern Hospital
Locations (1):
- Pamela Youde Nethersole Eastern Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No